CLINICAL TRIAL: NCT00902837
Title: Randomised, Double-blind, Double-dummy, Parallel-group Multicentre Study to Demonstrate Non-inferiority in Pain & Locomotor Function & Improvement in Symptoms of Constipation in Subjects With Moderate to Severe Pain Due to Osteoarthritis (OA) of the Knee &/or Hip Taking Oxycodone Equivalent of 20 - 80 mg/Day as Oxycodone/Naloxone Prolonged Release (OXN PR) Compared to Subjects Taking Oxycodone Prolonged Release Tablets (OxyPR) Alone.
Brief Title: OXN PR Compared to OxyPR to Demonstrate Non-inferiority in Pain & Locomotor Function & Improvement in Symptoms of Constipation in OA Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OXN3503; 2008-002670-36
Record Dates: First submitted 2009-05-14; First posted 2009-05-15 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Chronic Osteoarthritis
Keywords: randomised; double-blind; double-dummy; parallel-group; non-inferiority; pain locomotor function; improvement in symptoms of constipation; moderate to severe pain due to osteoarthritis (OA); OXN PR; OxyPR; Moderate to severe chronic nonmalignant OA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- oxycodone Tablet (Active Comparator): OxyCodone Prolonged release tablets
  Interventions: Drug: oxycodone prolonged release tablet
- oxycodone naloxone tablet (Experimental): Oxycodone naloxone prolonged release tablets (OXN)
  Interventions: Drug: Oxycodone naloxone prolonged release tablets (OXN); Drug: oxycodone naloxone tablet

INTERVENTIONS:
Drug: Oxycodone naloxone prolonged release tablets (OXN)
  Arms: oxycodone naloxone tablet
Drug: oxycodone prolonged release tablet
  Arms: oxycodone Tablet
Drug: oxycodone naloxone tablet
  Arms: oxycodone naloxone tablet

SUMMARY:
The primary objectives are

* to demonstrate that the treatment with OXN PR tablets is non-inferior to the treatment with OxyPR with regards to analgesic efficacy and locomotor function.
* to demonstrate that subjects with moderate to severe OA pain taking oxycodone/naloxone prolonged release tablets have improvement in symptoms of constipation compared to subjects taking oxycodone prolonged release tablets alone

DETAILED DESCRIPTION:
Subjects with moderate to severe pain due to osteoarthritis (OA) will be randomised to oxycodone/naloxone prolonged release (OXN PR) or oxycodone prolonged release tablets (OxyPR) alone to demonstrate that the treatment with OXN PR tablets is non-inferior to the treatment with OxyPR with regards to analgesic efficacy and locomotor function and to demonstrate that subjects taking OXN PR have improvement in symptoms of constipation compared to subjects taking OxyPR alone.

ELIGIBILITY:
Inclusion criteria:

* Moderate to severe chronic nonmalignant OA and that require around-the-clock opioid therapy.

Exclusion criteria:

* Females who are pregnant or lactating.
* Subjects with evidence of significant structural abnormalities of the gastrointestinal tract.
* Subjects with evidence of impaired liver/kidney function upon entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2009-05; Primary Completion 2010-04 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To demonstrate that treatment with OXN PR tablets is non-inferior to treatment with OxyPR with regards to analgesic efficacy & locomotor function. To demonstrate that subjects with moderate to severe OA pain taking oxycodone/naloxone prolonged re | End of 12 week study

CONTACTS AND LOCATIONS:
Locations (35):
- Ghent, Belgium
- Czechia (14):
  - Dr R Flasar, Brno
  - FN U Svate Anny, Brno
  - Urazova nemocnice v Brne, Brno
  - Dr E Lengalove, České Budějovice
  - Dr M Vdoviak, Karlovy Vary
  - Nemocnice Most, Most
  - Fakultni nemocnice Olomouc, Olomouc
  - Plzen-Lochotin
  - Revmatologicka ambulance, Prague
  - VFN Praha, Prague
  - Dr Z Urbanova, Prague
  - Chirurgicke oddeleni, Prague
  - FN Na Bulovce, Prague
  - Revmatologicka ambul, Uherské Hradiště
- Kuopio, Finland
- Germany (17):
  - Dr I Palutke, Bad Klosterlausnitz
  - Dr G Voss, Berlin
  - Schmerzzentrum Celle, Celle
  - Dr S Grunert, Eichstätt
  - Gemeinschaftspraxis fuer, Greifswald
  - Clinical Research, Hamburg
  - Praxis fur klinische Studien, Hamburg
  - Dr E A Lux, Lünen
  - Dr O Lowenstein, Mainz
  - Dr U Schutter, Marl
  - Dr H M Frick, Rhaunen
  - Prof Dr F Weber, Senftenberg
  - Senftenberg
  - Dr U Krauspe, Weimar
  - Dr J Hafer, Wetzlar
  - Intermed Institue fur Medizinische Forschung & Arzneimittelsicherheit, Wiesbaden
  - Schmerz und Palliativzentrum, Wiesbaden
- Mezőkövesd, Hungary
- Madrid, Spain

REFERENCES:
- See also: Text results available on website — https://www.clinicaltrialsregister.eu/ctr-search/search?query=OXN3503